CLINICAL TRIAL: NCT07169045
Title: Examination of the Validity and Reliability of 6-minute Stepper Test in Patients With Peripheral Artery Disease
Brief Title: Validity and Reliability of the 6-minute Stepper Test in Patients With Peripheral Artery Disease
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Study director, PT, PhD, Prof.Dr. Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Head of Cardiopulmonary Rehabilitation Clinic, Gazi University
Other Study IDs: 2025 - 1240
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Artery Disease (PAD)
Keywords: Peripheral Artery Disease; Exercise Testing; Validity and Reliability
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients With Peripheral Artery Disease

SUMMARY:
Hemodynamic dysfunction and decreased blood flow to the extremities negatively affect patients' muscle oxygenation, balance, claudication pain, lower extremity muscle strength, and arterial stiffness. These negatively affect patients' exercise capacity. The six-minute stepper test (6 MST) is a simple, low-cost, and minimal space requirement assessment method used to evaluate functional exercise capacity and is known to be valid and reliable for various pulmonary and cardiovascular diseases. However, it is not known whether the 6 MST is valid and reliable in assessing functional exercise capacity in patients with PAD. It is known that muscle oxygen levels, balance levels, intermittent claudication, lower extremity muscle strength, and arterial stiffness have negative effects on exercise capacity. However, the extent to which these variables affect the 6 MST is unknown. The primary aim is to examine the validity and reliability of the 6 MST in patients with PAD. The secondary aim is to evaluate arterial stiffness, muscle oxygen levels, intermittent claudication, static and dynamic balance levels, lower extremity muscle strength, and examine their effects on the 6 MST.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a common condition that carries a high risk of cardiovascular morbidity and mortality. PAD is an atherosclerotic process that causes occlusion of peripheral arteries. Hemodynamic dysfunction and decreased blood flow to the extremities negatively affect patients' muscle oxygenation, balance, claudication pain, lower extremity muscle strength, and arterial stiffness. These negatively affect patients' exercise capacity and increase the risk of mortality. To prevent this, patients' exercise capacity should be properly assessed and increased with an appropriate exercise programme. Several tests are available to assess exercise capacity. The cardiopulmonary exercise test (CPET) is the gold standard method for measuring exercise capacity. However, due to its high cost, the need for qualified personnel and complex equipment, it cannot be used in every clinic. Therefore, field tests have been developed to assess functional exercise capacity. The six-minute stepper test (6 MST) is a simple, low-cost, and minimal space requirement assessment method used to evaluate functional exercise capacity and is known to be valid and reliable for various pulmonary and cardiovascular diseases. However, it is not known whether the 6 MST is valid and reliable in assessing functional exercise capacity in patients with PAD. It is known that muscle oxygen levels, balance levels, intermittent claudication, lower extremity muscle strength, and arterial stiffness have negative effects on exercise capacity. However, the extent to which these variables affect the 6 MST is unknown. If this is known, clinicians and researchers will interpret this exercise test more carefully, and its use in individuals with PAD will become more effective. Therefore, the primary aim is to examine the validity and reliability of the 6 MST in patients with PAD. The secondary aim is to evaluate arterial stiffness, muscle oxygen levels, intermittent claudication, static and dynamic balance levels, lower extremity muscle strength, and examine their effects on the 6 MST. A minimum of 24 individuals with PAD will be included in the study. Patients' demographic and clinical information will be recorded. Pulmonary function (spirometry), PAD classification (Fonteine classification and Rutherford classification), and comorbidity (Charlson Comorbidity Index) will be assessed and recorded. The gold standard methods for assessing exercise capacity for structural validity, CPET and the 6-minute walk test (6 MWT), will be performed. For reliability, 6 MST will administered a second time at 24-hour intervals. Arterial stiffness (pulse wave analysis and brachial and aortic pulse wave velocity), muscle oxygenation (near-infrared spectrometer), peripheral muscle strength (dynamometer), static balance (Kinvent PLATES v3), dynamic balance (timed up and go test), intermittent claudication (Walking Impairment Questionnaire and Borg Scale) will assessed. The results will be analysed and interpreted using appropriate statistical analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with peripheral artery disease by the Department of Cardiovascular Surgery,
* Ankle-brachial index (ABI) ≤1.40 or exercise ABI ≤0.73 or diagnosed with calcified vascular response, in remission and under follow-up,
* Stable,
* Ages between 18 and 80,
* Patients who volunteer to participate in the study will be included.

Exclusion Criteria:

* Patients will be excluded if they have:
* Previously underwent ischaemic amputation,
* Unstable coronary artery disease,
* Uncontrolled Diabetes Mellitus,
* Pulmonary disease,
* Acute infection,
* Weight >110 kg because it is the upper limit of the stepper device,
* Contraindications to exercise testing per the American Sports Medicine Association,
* Pregnant and breastfeeding women,
* Patients with PAD who have undergone major surgery or had a myocardial infarction within the last 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 24 patients diagnosed with peripheral artery disease will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
6-minute Stepper Test | Trough study completion, an average of 1 year
  The test will performed using the previously defined Borel et al. criteria and the adaptation of the ATS/ERS 6 MWT criteria. For the test, a standard resistance 'Stepper' device will used, positioned 20 cm above the ground. To enable the patient to receive support if they lose their balance, the stepper device will placed 10 cm away from a straight wall edge. Patients will asked to take as many steps as possible during 6 minutes. The test will be conducted for 2 minutes first for the patient to learn, and then 6 minutes of testing will be conducted after a 3-minute rest period. 6 MST will be re-applied to patients 24 hours later using the same protocol for reliability analysis.
Cardiopulmonary Exercise Test | Trough study completion, an average of 1 year
  CPET is the gold standard method used to assess maximal exercise capacity. For this reason, 6 MST will used to examine structural validity. CPET will be performed using a gradually increasing workload protocol with breath-by-breath measurement on a treadmill. Electrocardiography (ECG) assessment during the test will be performed using a 12-lead ECG trace. Oxygen consumption and metabolic equivalent will be measured.
6-minute Walk Test | Trough study completion, an average of 1 year
  The 6 MWT is a valid and reliable submaximal exercise test for patients with peripheral arterial disease. 6 MWT will be applied to examine the structural validity of 6 MST. It will be carried out in accordance with ATS criteria.The walking distance will be recorded in two ways: in metres and as a percentage of the expected walking distance.

SECONDARY OUTCOMES:
Pulmonary function test | Trough study completion, an average of 1 year
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to American Thoracic Society and European Respiratory Society criteria. With the device, forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), FEV1/FVC, peak expiratory flow rate (PEF), and flow rate 25-75% of forced expiratory volume (FEV25-75%) will be measured.
Classification Systems for Peripheral Artery Disease | Trough study completion, an average of 1 year
  It will be performed using the Fontaine and Rutherford classification systems. According to the Fontaine classification system, peripheral arterial disease in individuals is assessed as stage I: asymptomatic disease, stage Ia: mild claudication, stage Ib: moderate-severe claudication, stage II: pain at rest, stage IV: ulceration or gangrene. According to the Rutherford classification system, it is classified as follows: 0: Asymptomatic, 1: Mild claudication, 2: Moderate claudication, 3: Severe claudication, 4: Ischemic rest pain, 5: Minor tissue loss, 6: Major tissue loss.
Charlson Comorbidity Index | Trough study completion, an average of 1 year
  This index identifies and defines 19 comorbid chronic diseases accompanying patients' primary diseases and determines the mortality risk. The total score obtained from the index ranges from 0 to 37.
Arterial Stiffness | Trough study completion, an average of 1 year
  Arterial stiffness will be assessed using the SphygmoCor® XCEL device. The patient's peripheral blood pressure will be measured by partially inflating the cuff on the brachial artery. Then, to assess carotid PWV, carotid pulse waves will be measured with a tonometer. A cuff will be placed on the femoral area to measure femoral PWV. The device will measure carotid-femoral artery PWV, pulse transit time, augmented index (Aix) values.
Peripheral Muscle Oxygenation | Trough study completion, an average of 1 year
  CPET and the second time applied 6 MST before, during, and recovery, the patients' dominant side gastrocnemius and quadriceps femoris muscles' oxygen percentage (SmO2%), oxyhaemoglobin (O2Hb) and deoxyhaemoglobin (HHb) levels, the difference between O2Hb and HHb (HbDiff), and total haemoglobin concentration (THb) levels will be measured using a near-infrared spectrometer (NIRS) device.
Peripheral Muscle Strength | Trough study completion, an average of 1 year
  Patients' knee extensor and plantar flexor muscle strength will be assessed using the Kinvent K-Push dynamometer.
Static Balance | Trough study completion, an average of 1 year
  Static balance assessment will be performed using Kinvent PLATES v3. On the PLATES, with eyes open and closed, three repetitions will be performed first on double leg and then single leg. The average of the three tests will be used for analysis.
Dynamic Balance | Trough study completion, an average of 1 year
  Dynamic balance will be assessed using the timed up and go test. The duration will be recorded in seconds. The test will be repeated three times, and the best time will be used in the analysis.
Walking Impairment Questionnaire (WIQ) | Trough study completion, an average of 1 year
  The 21-item 'Walking Impairment Questionnaire (WIQ)' developed by Regensteiner et al. (1995) will be used in its Turkish adaptation. WIQ consists of the parameters of claudication, differential diagnosis, walking distance, walking speed, and the ability to climb stairs. A high score indicates high performance.
Intermittent Claudication | Trough study completion, an average of 1 year
  Intermittent claudication will recorded using the modified Borg scale. The total number of steps at the end of the 6 MST, the time when claudication pain began, the number of steps at which claudication pain began, the duration of the test in minutes, and whether absolute claudication pain was present will recorded. The onset time and distance of intermittent claudication and absolute claudication will be recorded in the CPET and 6 MWT tests.
Dyspnea Perception | Trough study completion, an average of 1 year
  Dyspnea perception will be measured with Modified Borg Scale. The Modified Borg scale is a subjective scale that scores 0-10 for breathlessness and fatigue at rest and/or during activity. The lowest 0 points "not at all" the highest 10 points "very severe" means shortness of breath. before, during, and after the The perception of dyspnea will be assessed before, during, and recovery of the 6 MST, CPET, and 6 MWT.
Fatigue Perception | Trough study completion, an average of 1 year
  Fatigue perception will be evaluated with Modified Borg Scale. The Modified Borg scale is a subjective scale that scores 0-10 for breathlessness and fatigue at rest and/or during activity. The lowest 0 points "not at all" the highest 10 points "very severe" means fatigue. The perception of fatigue will be assessed before, during, and recovery of the 6 MST, CPET, and 6 MWT.

CONTACTS AND LOCATIONS:
Overall Officials: Beyza BEKDEMİR, Study Chair — Gazi University; Nihan KATAYIFÇI, Principal Investigator — Gazi University; Abdullah ÖZER, Principal Investigator — Gazi University; Meral BOŞNAK GÜÇLÜ, Study Director — Gazi University
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schieber MN, Hasenkamp RM, Pipinos II, Johanning JM, Stergiou N, DeSpiegelaere HK, Chien JH, Myers SA. Muscle strength and control characteristics are altered by peripheral artery disease. J Vasc Surg. 2017 Jul;66(1):178-186.e12. doi: 10.1016/j.jvs.2017.01.051. PMID 28647034
- [Background] Gohil RA, Mockford KA, Mazari F, Khan J, Vanicek N, Chetter IC, Coughlin PA. Balance impairment, physical ability, and its link with disease severity in patients with intermittent claudication. Ann Vasc Surg. 2013 Jan;27(1):68-74. doi: 10.1016/j.avsg.2012.05.005. Epub 2012 Oct 18. PMID 23084732
- [Result] Parmenter BJ, Dieberg G, Smart NA. Exercise training for management of peripheral arterial disease: a systematic review and meta-analysis. Sports Med. 2015 Feb;45(2):231-44. doi: 10.1007/s40279-014-0261-z. PMID 25230780
- [Result] Collins EG, McBurney C, Butler J, Jelinek C, O'Connell S, Fritschi C, Reda D. The Effects of Walking or Walking-with-Poles Training on Tissue Oxygenation in Patients with Peripheral Arterial Disease. Int J Vasc Med. 2012;2012:985025. doi: 10.1155/2012/985025. Epub 2012 Sep 25. PMID 23050152
- [Result] Catalano M, Scandale G, Carzaniga G, Cinquini M, Minola M, Dimitrov G, Carotta M. Increased aortic stiffness and related factors in patients with peripheral arterial disease. J Clin Hypertens (Greenwich). 2013 Oct;15(10):712-6. doi: 10.1111/jch.12167. Epub 2013 Jul 16. PMID 24088278
- [Result] Durukan BN, Ozcan EB, Saglam M, Sener YZ, Vardar-Yagli N, Ince DI, Tokgozoglu L, Calik-Kutukcu E. Validity and reliability of the 6-min stepper test in hypertensive individuals. J Hypertens. 2025 May 1;43(5):880-886. doi: 10.1097/HJH.0000000000003996. Epub 2025 Mar 5. PMID 40079829
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Result] Borel B, Fabre C, Saison S, Bart F, Grosbois JM. An original field evaluation test for chronic obstructive pulmonary disease population: the six-minute stepper test. Clin Rehabil. 2010 Jan;24(1):82-93. doi: 10.1177/0269215509343848. PMID 20053721
- [Result] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I; ESC Scientific Document Group. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS): Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteriesEndorsed by: the European Stroke Organization (ESO)The Task Force for the Diagnosis and Treatment of Peripheral Arterial Diseases of the European Society of Cardiology (ESC) and of the European Society for Vascular Surgery (ESVS). Eur Heart J. 2018 Mar 1;39(9):763-816. doi: 10.1093/eurheartj/ehx095. No abstract available. PMID 28886620